CLINICAL TRIAL: NCT03977155
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of BOS-589 in the Treatment of Patients With Diarrhea-predominant Irritable Bowel Syndrome (IBS-D)
Brief Title: Study to Evaluate the Efficacy, Safety, and Tolerability of BOS-589 in the Treatment of Patients With Diarrhea-predominant Irritable Bowel Syndrome (IBS-D)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BOS-589-201
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Diarrhea-predominant Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; diarrhea; BOS-589
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High dose of BOS-589 (Experimental): Participants will receive a high dose of BOS-589 orally twice a day (BID).
  Interventions: Drug: BOS-589
- Low dose of BOS-589 (Experimental): Participants will receive a low dose of BOS-589 orally BID.
  Interventions: Drug: BOS-589
- Placebo (Placebo Comparator): Participants will receive matching placebo orally BID.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BOS-589 — oral tablets
  Arms: High dose of BOS-589; Low dose of BOS-589
Drug: Placebo — oral tablets
  Arms: Placebo

SUMMARY:
This study is being conducted to evaluate in participants with diarrhea-predominant Irritable Bowel Syndrome (IBS-D) the abdominal pain response to BOS-589 after 4 weeks of treatment and to evaluate the overall safety and tolerability of BOS-589 in the treatment of IBS-D during 4 weeks of treatment, relative to placebo (PBO).

ELIGIBILITY:
Inclusion Criteria:

* Participant meets the diagnosis of diarrhea-predominant IBS (IBS-D) subtype based on Rome IV diagnostic criteria within 3 months prior to randomization. On days when the participant experiences IBS symptoms

  * At least 25% of stools are loose or watery; and
  * Fewer than 25% of stools are hard.
* Recurrent abdominal pain occurring, on average, at least 1 day per week and associated with 2 or more of the following:

  * Related to defecation;
  * Associated with a change in frequency of bowel movements;
  * Associated with a change in form (appearance) of stool.
* Over the week prior to randomization, the participant has

  * An average of worst abdominal pain (WAP) scores in the prior 24 hours of 4.0 to 8.0 on a 0 to 10 numerical rating scale;
  * An average daily Bristol Stool Form Scale (BSFS) score ≥ 5.0 (and at least 5 days with a BSFS score ≥ 5.0;
  * An average daily IBS-Global Scale (IBS-GS) score of ≥ 2.0.
* Participant must undergo or previously have undergone (a) an appropriate evaluation for their IBS symptoms, including an evaluation for organic/structural etiologies (if in the presence of alarm symptoms); and (b) age-appropriate screening for colorectal cancer, if applicable.
* Participant is negative for serum tissue transglutaminase immunoglobulin A antibody (tTG-IgA) plus has evidence of detectable serum IgA within the normal reference range.

Exclusion Criteria:

* At the time of screening, participant has a diagnosis of an IBS subtype other than IBS-D, based on Rome IV criteria.
* Participant has a history of inflammatory or immune-mediated gastrointestinal (GI) disorders including (but not limited to) inflammatory bowel disease (i.e., Crohn's disease, ulcerative colitis, microscopic colitis, and celiac disease).
* Participant has had an episode of diverticulitis within 3 months prior to Screening.
* Participant has a history of intestinal obstruction, stricture, toxic megacolon, GI perforation, fecal impaction, gastric banding, bariatric surgery, adhesions, ischemic colitis, or impaired intestinal circulation (e.g., aortoiliac occlusive disease).
* Participant has any of the following surgical history:

  * Cholecystectomy with any history of post-cholecystectomy biliary tract pain;
  * Any abdominal surgery within the 3 months prior to Screening;
  * Major gastric, esophageal, hepatic, pancreatic, or intestinal surgery (appendectomy, hemorrhoidectomy, or polypectomy greater than 3 months post-surgery are allowed).
* Confirmed alanine aminotransferase (ALT) > 2 upper limit of normal (ULN)
* Confirmed total bilirubin > ULN, unless the participant has a documented history of Gilbert's syndrome
* Evidence of active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection or Human immunodeficiency virus (HIV)-1 or HIV-2 antibody positive
* Evidence of HCV infection based on a positive HCV antibody screen (Participants who have been successfully treated for HCV are eligible if an undetectable HCV viral load at least 6 months after completion of treatment can be demonstrated.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (58):
- United States (58):
  - Pinnacle Research Group, Anniston, Alabama
  - Clinical Research Associates, Huntsville, Alabama
  - Synexus Clinical Research US, Inc. - East Valley Family Physicians, PLC, Chandler, Arizona
  - Synexus Clinical Research US, Inc. - Phoenix Southeast, Chandler, Arizona
  - Synexus Clinical Research US, Inc. - Desert Clinical Research, LLC, Mesa, Arizona
  - Synexus Clinical Research US, Inc. - Central Arizona Medical Associates, PC, Mesa, Arizona
  - Hope Research Institute LLC, Peoria, Arizona
  - Elite Clinical Studies, Phoenix, Arizona
  - Synexus Clinical Research US, Inc. - Tatum Highlands Medical Associates, PLLC, Phoenix, Arizona
  - Hope Research Institute LLC, Phoenix, Arizona
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Synexus Clinical Research US, Inc., Carlsbad, California
  - Paragon Rx Clinical, Inc., Garden Grove, California
  - eStudySite, La Mesa, California
  - Grossmont Center For Clinical Research, La Mesa, California
  - Clinical Trials Research, Sacramento, California
  - Research and Education Inc, San Diego, California
  - Precision Research Institute, San Diego, California
  - Shahram Jacobs MD Inc, Sherman Oaks, California
  - Millennium ClinicalTrials, Thousand Oaks, California
  - Advanced Rx Clinical Research, Westminster, California
  - Chase Medical Research LLC, Waterbury, Connecticut
  - PAB Clinical Research-ClinEdge-PPDS, Brandon, Florida
  - Nature Coast Clinical Research LLC - ERN-PPDS, Inverness, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Health Awareness Inc, Jupiter, Florida
  - Suncoast Research Group LLC - ERN-PPDS, Miami, Florida
  - Ormond Medical Arts Pharmaceutical, Ormond Beach, Florida
  - Precision Clinical Research, LLC, Sunrise, Florida
  - Northwest Clinical Trials-ClinEdge-PPDS, Boise, Idaho
  - Synexus Clinical Research US, Inc. - Allaw, Evansville, Indiana
  - Boston Clinical Trials Inc, Boston, Massachusetts
  - West Michigan Clinical Research, Wyoming, Michigan
  - Sundance Clinical Research, St Louis, Missouri
  - Quality Clinical Research - ClinEdge - PPDS, Omaha, Nebraska
  - Albuquerque Clinical Trials Inc - BTC - PPDS, Albuquerque, New Mexico
  - NY Scientific, Brooklyn, New York
  - Peters Medical Research, LLC, High Point, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - Synexus Clinical Research US, Inc., Akron, Ohio
  - Hometown Urgent Care and Research, Cincinnati, Ohio
  - Synexus Clinical Research US, Inc., Columbus, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - Founders Research Corporation, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Safe Harbor Clinical Research, East Providence, Rhode Island
  - Synexus Clinical Research US, Inc., Anderson, South Carolina
  - Pledmont Research Partners LLC, Fort Mill, South Carolina
  - Synexus Clinical Research US, Inc., Greer, South Carolina
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - New Phase Research & Development, Knoxville, Tennessee
  - L12 Clinical Research, Dallas, Texas
  - Synexus Clinical Research US, Inc., Dallas, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Quality Research Inc., San Antonio, Texas
  - Advanced Research Institute, Ogden, Utah
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Clinical Research Partners LLC, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 47 study centers in the United States.
Pre-assignment Details: During the pretreatment phase, participants were evaluated for up to 5 weeks to assess eligibility. The pretreatment phase consisted of initial screening assessments and a run in period.
Groups:
- High Dose of BOS-589: Randomized participants received a high dose of BOS-589 tablets orally twice a day (BID).
- Low Dose of BOS-589: Randomized participants received a low dose of BOS-589 tablets orally BID.
- Placebo: Randomized participants received matching placebo tablets orally BID.
Period: Overall Study
Arm/Group | High Dose of BOS-589 | Low Dose of BOS-589 | Placebo
Started | 43 | 48 | 42
Completed | 38 | 46 | 40
Not Completed | 5 | 2 | 2
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Participant was unable to come in for the Visit | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- High Dose of BOS-589: Randomized participants received a high dose of BOS-589 tablets orally BID.
- Total: Total of all reporting groups
Arm/Group | High Dose of BOS-589 | Low Dose of BOS-589 | Placebo | Total
Number analyzed (Participants) | 43 | 48 | 42 | 133
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.0 (13.15) | 39.9 (13.26) | 40.0 (12.84) | 40.3 (13.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 26 | 87
  Male | 13 | 17 | 16 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 7 | 20
  Not Hispanic or Latino | 37 | 41 | 35 | 113
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 3 | 7 | 6 | 16
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 2 | 8 | 2 | 12
  White | 36 | 33 | 34 | 103
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 24-hour Worst Abdominal Pain Scores (WAP) at Day 29 Compared to Baseline (Averaged Over the Week Prior to Each Respective Time Point)
Description: To evaluate in participants with diarrhea-predominant irritable bowel syndrome (IBS-D) the abdominal pain response to BOS-589 after 4 weeks of treatment, relative to placebo. Throughout the 4 weeks of the double blind treatment phase, participants were asked to rate their WAP in the past 24 hours. The participant-reported WAP in the past 24 hours was recorded on a 0 to 10 scale, where 0 corresponded to no pain and 10 corresponded to worst imaginable pain. Higher scores indicated worse outcome.
Time Frame: Baseline; Day 29
Population: The Intent to Treat (ITT) Analysis Set included all randomized participants. Here, overall number of participants analyzed signifies only the participants with available data that were analyzed for the outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- BOS-589: Active Treatment: High Dose of BOS-589: Randomized participants received a high dose of BOS-589 tablets orally BID.
  Low Dose of BOS-589: Randomized participants received a low dose of BOS-589 tablets orally BID.
  Data were pooled from the above mentioned doses for analysis.
Arm/Group | High Dose of BOS-589 | Low Dose of BOS-589 | BOS-589: Active Treatment | Placebo
Number analyzed (Participants) | 39 | 46 | 85 | 40
Score on a scale | -1.64 (1.684) | -2.30 (1.933) | -2.00 (1.842) | -1.69 (1.783)
Statistical Analysis 1: Comparison: BOS-589: Active Treatment vs Placebo; Statistical Analysis 1; Test type: Superiority — Individual BOS-589 dose levels versus placebo were only to be tested if pooled BOS-589 doses versus placebo was significant at p<0.05; p = 0.3776, t test; P-values were calculated from the independent two-sample t test with equal variance; Mean Difference (Net) = -0.31, 95% CI 2-sided [-1.00 to 0.38], Standard Error of Mean 0.350
Statistical Analysis 2: Comparison: High Dose of BOS-589 vs Placebo; Statistical Analysis 2; Test type: Superiority; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.73 to 0.82], Standard Error of Mean 0.390
Statistical Analysis 3: Comparison: Low Dose of BOS-589 vs Placebo; Statistical Analysis 3; Test type: Superiority; Mean Difference (Net) = -0.61, 95% CI 2-sided [-1.41 to 0.19], Standard Error of Mean 0.403
Statistical Analysis 4: Comparison: High Dose of BOS-589 vs Low Dose of BOS-589; Statistical Analysis 4; Test type: Superiority; Mean Difference (Net) = 0.65, 95% CI 2-sided [-0.13 to 1.44], Standard Error of Mean 0.397

2. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Discontinuations Because of AEs, and Any Treatment-related Severe AEs
Description: To evaluate the overall safety and tolerability of BOS-589 in the treatment of IBS-D during 4 weeks of treatment, relative to placebo.
Time Frame: Up to Day 43/end-of-study follow up visit
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | High Dose of BOS-589 | Low Dose of BOS-589 | Placebo
Number analyzed (Participants) | 43 | 48 | 42
Participants
  Any Treatment-emergent adverse event (TEAE) | 23 | 23 | 15
  Any TEAE Related to Study Drug | 8 | 5 | 4
  Any Moderate or Severe TEAE | 10 | 10 | 6
  Any Moderate or Severe TEAE Related to Study Drug | 3 | 3 | 1
  Any Treatment-Emergent SAE | 0 | 0 | 0
  Any Treatment-Emergent SAE Related to Study Drug | 0 | 0 | 0
  Any TEAE Causing Discontinuation of Study Drug | 3 | 0 | 0
  Any TEAE Leading to Withdrawal from the Study | 3 | 0 | 0
  Any TEAE with Outcome of Death | 0 | 0 | 0

3. Secondary Outcome: Change in Stool Consistency, Measured by the Daily Bristol Stool Form Score (BSFS) Most Representative Stool Consistency Scores at Day 29 Compared to Baseline (Averaged Over the Week Prior to Each Respective Time Point)
Description: To evaluate the treatment effect of BOS-589 on defecation after 4 weeks, relative to placebo. Participants were asked to record daily stool consistency according to the BSFS most representative of the past 24 hours. The participant-reported BSFS consistency score was based on a 1 to 7 scale where 1 corresponded to a hard stool and 7 corresponded to watery diarrhea. Higher scores indicated worse outcome.
Time Frame: Baseline; Day 29
Population: The ITT Analysis Set included all randomized participants. Here, overall number of participants analyzed signifies only the participants with available data that were analyzed for the outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | High Dose of BOS-589 | Low Dose of BOS-589 | BOS-589: Active Treatment | Placebo
Number analyzed (Participants) | 39 | 45 | 84 | 40
Score on a scale | -1.11 (1.179) | -0.97 (1.087) | -1.04 (1.125) | -1.01 (1.034)
Statistical Analysis 1: Comparison: BOS-589: Active Treatment vs Placebo; Statistical Analysis 1; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.8840, t test; P-values were calculated from the independent two-sample t test with equal variance; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.45 to 0.39], Standard Error of Mean 0.211
Statistical Analysis 2: Comparison: High Dose of BOS-589 vs Placebo; Statistical Analysis 2; Test type: Superiority; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.60 to 0.39], Standard Error of Mean 0.249
Statistical Analysis 3: Comparison: Low Dose of BOS-589 vs Placebo; Statistical Analysis 3; Test type: Superiority; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.43 to 0.49], Standard Error of Mean 0.231
Statistical Analysis 4: Comparison: High Dose of BOS-589 vs Low Dose of BOS-589; Statistical Analysis 4; Test type: Superiority; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.63 to 0.36], Standard Error of Mean 0.247

4. Secondary Outcome: Change in Stool Consistency, Measured by the Daily BSFS Worst (Loosest) Stool Consistency Scores at Day 29 Compared to Baseline (Averaged Over the Week Prior to Each Respective Time Point)
Description: To evaluate the treatment effect of BOS-589 on defecation after 4 weeks, relative to placebo. Participants were asked to record daily stool consistency according to the BSFS worst stool consistency (defined as the loosest stool with the highest BSFS score) in the past 24 hours. The participant-reported BSFS consistency score was based on a 1 to 7 scale where 1 corresponded to a hard stool and 7 corresponded to watery diarrhea. Higher scores indicated worse outcome.
Time Frame: Baseline; Day 29
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | High Dose of BOS-589 | Low Dose of BOS-589 | BOS-589: Active Treatment | Placebo
Number analyzed (Participants) | 37 | 40 | 77 | 32
Score on a scale | -1.13 (1.167) | -1.06 (1.132) | -1.09 (1.142) | -0.93 (0.926)
Statistical Analysis 1: Comparison: BOS-589: Active Treatment vs Placebo; Statistical Analysis 1; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.4725, t test; P-values were calculated from the independent two-sample t test with equal variance; Mean Difference (Net) = -0.16, 95% CI 2-sided [-0.62 to 0.29], Standard Error of Mean 0.228
Statistical Analysis 2: Comparison: High Dose of BOS-589 vs Placebo; Statistical Analysis 2; Test type: Superiority; Median Difference (Final Values) = -0.20, 95% CI 2-sided [-0.71 to 0.31], Standard Error of Mean 0.256
Statistical Analysis 3: Comparison: Low Dose of BOS-589 vs Placebo; Statistical Analysis 3; Test type: Superiority; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.62 to 0.37], Standard Error of Mean 0.248
Statistical Analysis 4: Comparison: High Dose of BOS-589 vs Low Dose of BOS-589; Statistical Analysis 4; Test type: Superiority; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.60 to 0.45], Standard Error of Mean 0.262

5. Secondary Outcome: Change in Stool Frequency, Measured by the Total Number of Spontaneous Bowel Movements in 24 Hours at Day 29 Compared to Baseline (Averaged Over the Week Prior to Each Respective Time Point)
Description: To evaluate the treatment effect of BOS-589 on defecation after 4 weeks, relative to placebo. Participants were asked to record stool frequency based on the total number of spontaneous bowel movements in the past 24 hours.
Time Frame: Baseline; Day 29
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Number of spontaneous bowel movements
Arm/Group | High Dose of BOS-589 | Low Dose of BOS-589 | BOS-589: Active Treatment | Placebo
Number analyzed (Participants) | 39 | 46 | 85 | 40
Number of spontaneous bowel movements | -0.69 (1.190) | -0.74 (0.944) | -0.71 (1.057) | -0.83 (1.006)
Statistical Analysis 1: Comparison: BOS-589: Active Treatment vs Placebo; Statistical Analysis 1; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.5693, t test; P-values were calculated from the independent two-sample t test with equal variance; Mean Difference (Net) = 0.11, 95% CI 2-sided [-0.28 to 0.51], Standard Error of Mean 0.200
Statistical Analysis 2: Comparison: High Dose of BOS-589 vs Placebo; Statistical Analysis 2; Test type: Superiority; Mean Difference (Net) = 0.14, 95% CI 2-sided [-0.35 to 0.63], Standard Error of Mean 0.248
Statistical Analysis 3: Comparison: Low Dose of BOS-589 vs Placebo; Statistical Analysis 3; Test type: Superiority; Mean Difference (Net) = 0.09, 95% CI 2-sided [-0.33 to 0.51], Standard Error of Mean 0.210
Statistical Analysis 4: Comparison: High Dose of BOS-589 vs Low Dose of BOS-589; Statistical Analysis 4; Test type: Superiority; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.41 to 0.51], Standard Error of Mean 0.231

6. Secondary Outcome: Changes in the Irritable Bowel Syndrome-Severity Score (IBS-SS) at Day 29 Compared to Baseline
Description: To evaluate the treatment effect of BOS-589 on IBS-related signs and symptoms. Participants were asked to complete 5 questions regarding the severity of their IBS. Each of the 5 questions generated a maximum score of 100, leading to a total possible IBS-SS of 500. The IBS-SS scale ranges from 0 to 500. A higher score indicated greater severity.
Time Frame: Baseline; Day 29
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | High Dose of BOS-589 | Low Dose of BOS-589 | BOS-589: Active Treatment | Placebo
Number analyzed (Participants) | 30 | 37 | 67 | 30
Score on a scale | -89.3 (116.65) | -146.8 (113.06) | -121.0 (117.38) | -113.3 (108.51)
Statistical Analysis 1: Comparison: BOS-589: Active Treatment vs Placebo; Statistical Analysis 1; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.7603, t test; P-values were calculated from the independent two-sample t test with equal variance; Mean Difference (Net) = -7.71, 95% CI 2-sided [-57.76 to 42.33], Standard Error of Mean 25.208
Statistical Analysis 2: Comparison: High Dose of BOS-589 vs Placebo; Statistical Analysis 2; Test type: Superiority; Mean Difference (Net) = 24.00, 95% CI 2-sided [-34.22 to 82.22], Standard Error of Mean 29.087
Statistical Analysis 3: Comparison: Low Dose of BOS-589 vs Placebo; Statistical Analysis 3; Test type: Superiority; Mean Difference (Net) = -33.42, 95% CI 2-sided [-87.91 to 21.07], Standard Error of Mean 27.285
Statistical Analysis 4: Comparison: High Dose of BOS-589 vs Low Dose of BOS-589; Statistical Analysis 4; Test type: Superiority; Mean Difference (Net) = 57.42, 95% CI 2-sided [1.16 to 113.69], Standard Error of Mean 28.174

7. Secondary Outcome: Change in the IBS Global Scale (IBS-GS) at Day 29 Compared to Baseline (Averaged Over the Week Prior to Each Respective Time Point)
Description: To evaluate the treatment effect of BOS-589 on IBS related signs and symptoms. Participants were asked to record daily their overall diarrhea-predominant Irritable Bowel Syndrome (IBS-D) global symptoms in the prior 24 hours. The participant-reported daily IBS-GS was based on a 0 to 4 scale where: 0 corresponded to no symptoms; 1 corresponded to mild symptoms; 2 corresponded to moderate symptoms; 3 corresponded to severe symptoms; and 4 corresponded to very severe symptoms. Higher scores indicated severe symptoms.
Time Frame: Baseline; Day 29
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | High Dose of BOS-589 | Low Dose of BOS-589 | BOS-589: Active Treatment | Placebo
Number analyzed (Participants) | 39 | 46 | 85 | 40
Score on a scale | -0.56 (0.629) | -0.89 (0.815) | -0.74 (0.750) | -0.57 (0.626)
Statistical Analysis 1: Comparison: BOS-589: Active Treatment vs Placebo; Statistical Analysis 1; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.2149, t test; P-values were calculated from the independent two-sample t test with equal variance; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.44 to 0.10], Standard Error of Mean 0.137
Statistical Analysis 2: Comparison: High Dose of BOS-589 vs Placebo; Statistical Analysis 2; Test type: Superiority; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.27 to 0.29], Standard Error of Mean 0.141
Statistical Analysis 3: Comparison: Low Dose of BOS-589 vs Placebo; Statistical Analysis 3; Test type: Superiority; Mean Difference (Net) = -0.32, 95% CI 2-sided [-0.64 to -0.01], Standard Error of Mean 0.159
Statistical Analysis 4: Comparison: High Dose of BOS-589 vs Low Dose of BOS-589; Statistical Analysis 4; Test type: Superiority; Mean Difference (Net) = 0.33, 95% CI 2-sided [0.02 to 0.65], Standard Error of Mean 0.160

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for BOS-589
Description: To evaluate the steady state pharmacokinetics (PK) of BOS-589.
Time Frame: Day 1, Day 15 and Day 22 at pre-dose and at 0.5, 1, 2, and 4 hours post-dose
Population: The PK population included all participants who took any amount of BOS-589 and had sufficient concentration time data to report at least a maximum concentration (Cmax). Here, number analyzed in each row signifies only the participants with available data that were analyzed for that day.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | High Dose of BOS-589 | Low Dose of BOS-589
Number analyzed (Participants) | 43 | 48
pg/mL
  Day 1: number analyzed (Participants) | 39 | 48
  Day 1 | 1840 (90.4) | 999 (72.0)
  Day 15: number analyzed (Participants) | 32 | 39
  Day 15 | 2050 (109) | 1280 (91.2)
  Day 22: number analyzed (Participants) | 5 | 5
  Day 22 | 984 (105) | 1620 (117)

9. Secondary Outcome: Time to Reach Cmax (Tmax) for BOS-589
Description: To evaluate the steady state PK of BOS-589.
Time Frame: Day 1, Day 15 and Day 22 at pre-dose and at 0.5, 1, 2, and 4 hours post-dose
Population: as for outcome 8
Measure: Median (Full Range); unit: Hour
Arm/Group | High Dose of BOS-589 | Low Dose of BOS-589
Number analyzed (Participants) | 43 | 48
Hour
  Day 1: number analyzed (Participants) | 39 | 48
  Day 1 | 1.02 [0.42 to 4.00] | 1.21 [0.50 to 4.05]
  Day 15: number analyzed (Participants) | 32 | 39
  Day 15 | 1.44 [0.50 to 4.02] | 1.05 [0.00 to 4.00]
  Day 22: number analyzed (Participants) | 5 | 5
  Day 22 | 1.00 [0.00 to 2.00] | 1.92 [1.92 to 2.03]

10. Secondary Outcome: Area Under the Concentration-versus-time Curve (AUC) From Time Zero to 4 Hours Post Dose (AUC0-4) for BOS-589
Description: To evaluate the steady state PK of BOS-589.
Time Frame: Day 1, Day 15 and Day 22 at pre-dose and at 0.5, 1, 2, and 4 hours post-dose
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | High Dose of BOS-589 | Low Dose of BOS-589
Number analyzed (Participants) | 43 | 48
h*pg/mL
  Day 1: number analyzed (Participants) | 38 | 45
  Day 1 | 4250 (90.5) | 2460 (65.3)
  Day 15: number analyzed (Participants) | 31 | 38
  Day 15 | 6080 (85.4) | 3090 (91.5)
  Day 22: number analyzed (Participants) | 4 | 4
  Day 22 | 2210 (85.9) | 7360 (38.9)

11. Secondary Outcome: AUC From Time Zero to the Last Quantifiable Concentration (AUC0-t) for BOS-589
Description: To evaluate the steady state PK of BOS-589.
Time Frame: Day 1, Day 15 and Day 22 at pre-dose and at 0.5, 1, 2, and 4 hours post-dose
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | High Dose of BOS-589 | Low Dose of BOS-589
Number analyzed (Participants) | 43 | 48
h*pg/mL
  Day 1: number analyzed (Participants) | 39 | 47
  Day 1 | 4330 (90.3) | 2470 (63.7)
  Day 15: number analyzed (Participants) | 31 | 39
  Day 15 | 6080 (85.4) | 3220 (96.9)
  Day 22: number analyzed (Participants) | 5 | 5
  Day 22 | 2480 (78.5) | 4640 (149)

ADVERSE EVENTS:
Time Frame: Up to Day 43/end-of-study follow up visit
Arm/Group | High Dose of BOS-589 | Low Dose of BOS-589 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/48 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/48 | 0/42
Other Adverse Events (participants affected / at risk) | 23/43 | 23/48 | 15/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose of BOS-589 (N=43) | Low Dose of BOS-589 (N=48) | Placebo (N=42)
Nasopharyngitis (Infections and infestations) | 2 | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 1
Urinary tract infection (Infections and infestations) | 2 | 2 | 0
Influenza (Infections and infestations) | 0 | 2 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 4 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 4 | 4
Dizziness (Nervous system disorders) | 2 | 1 | 2
Migraine (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 1
Post procedural contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Catheter site bruise (General disorders) | 1 | 0 | 1
Catheter site pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0
Red blood cell sedimentation rate increased (Investigations) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT03977155/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT03977155/SAP_001.pdf